CLINICAL TRIAL: NCT00804921
Title: Effectiveness of Oral Acetazolamide, Brimonidine Tartarate, and Anterior Chamber Paracentesis for Ocular Hypertension Control After Intravitreal Bevacizumab Injection: Preliminary Results
Brief Title: Effectiveness of Oral Acetazolamide, Brimonidine Tartarate, and Anterior Chamber Paracentesis in Intraocular Pressure (IOP) After Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: CONEP (Comite Nacional de Etica em Pesquisa)
Other Study IDs: IOP After Bevacizumab
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Macular Edema; Diabetic Retinopathy; Macular Degeneration
Keywords: bevacizumab; intra-ocular pressure; acetazolamide; anterior chamber paracentesis; brimonidine; macular edema secondary to diabetic retinopathy or macular degeneration
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy; Macular Degeneration | interventions — Bevacizumab; Acetazolamide; Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bevacizumab
Procedure: anterior chamber paracentesis
Drug: acetazolamide
Drug: brimonidine

SUMMARY:
Purpose: To evaluate the effects of anterior chamber paracentesis, brimonidine and oral acetazolamide to reduce intra-ocular pressure (IOP) variations after intravitreal bevacizumab injection (IVBV).

Methods: 47 patients scheduled for IVBV (1.5 mg / 0.06 ml) will be randomly assigned to a pre-treatment 1 hour before IVBV with either 250 mg oral acetazolamide (DIA, 9 eyes), anterior chamber paracentesis immediate after IVBV (PAR, 15 eyes), topic brimonidine tartarate 1 hour before IVBV (BRI, 14 eyes), or no pre-treatment IBVB (CTR, 9 eyes). IOP will be measured 90 minutes before injection (baseline), just before injection, and at 3, 10, 20 and 30 minutes after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* macular edema

Exclusion Criteria:

* pulmonary chronic problems
* chronic renal failure
* intraocular inflammation
* drug or alcohol addiction

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Intra-ocular pressure variation after intra-vitreous injection of bevacizumab

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine - Clinical Hospital, Ribeirão Preto, São Paulo, Brazil